CLINICAL TRIAL: NCT05927753
Title: A Randomized, Active-Controlled, Open-Label Study to Evaluate the Clinical Performance of Deseyne (Vifilcon C) Daily Disposable Soft Contact Lens
Brief Title: Study to Evaluate the Clinical Performance of Deseyne (Vifilcon C) Daily Disposable Soft Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruno Vision Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BrunoVisionCare22001
Record Dates: First submitted 2023-05-31; First posted 2023-07-03 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2023-06

CONDITIONS: Refractive Error - Myopia Bilateral

STUDY DESIGN:
Intervention Model Description: Comparison of a test contact lens performance to a known, cleared for market contact lens.
Masking Description: Open label randomization assignment between test and control intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Test lens. Deseyne Daily Disposable Contact Lens (Experimental): Test contact lens to be worn as a daily disposable soft (hydrophilic) contact lens, to be discarded daily. Individual new lens placed daily for a period of 90 consecutive days, bilaterally. Follow-up visits are 1 week, 1 month, 2 months, and 3 months after dispensing.
  Interventions: Device: Deseyne Daily Disposable Contact Lens (Test Device)
- Control lens. 1-Day Acuvue Moist Daily Disposable Contact Lens (Active Comparator): Control lens to be worn as a daily disposable soft (hydrophilic) contact lens, to be discarded daily, Individual new lens placed daily for a period of 90 consecutive days, bilaterally. Follow-up visits are 1 week, 1 month, 2 months, and 3 months after dispensing.
  Interventions: Device: Deseyne Daily Disposable Contact Lens (Test Device)

INTERVENTIONS:
Device: Deseyne Daily Disposable Contact Lens (Test Device) — Comparison of contact lens performance between the test lens under study (Deseyne Daily Disposable Contact Lens) and the control lens f(1-Day Acuvue Moist Contact Lens) for safety and effectiveness.

SUMMARY:
This clinical study is to provide clinical performance data comparing the test lens (Deseyne [vifilcon C] daily disposable soft contact lens) to a control lens (1-Day Acuvue Moist [etafilcon A] daily disposable soft contact lens) in the same indication for use (single use prior to removal followed by a fresh lens upon the next lens wear exposure). The study is designed to test the hypothesis that the test lens is substantially equivalent to the control lens in like indications for use.

DETAILED DESCRIPTION:
A multicenter, randomized, active-controlled, open-label study design will be used to compare the clinical performance of the Deseyne (vifilcon C) test soft contact lens to the similarly indicated 1-Day Acuvue® Moist® (etafilcon A) control soft contact lens.

Study participation is approximately 90 days in duration and will consist of approximately 80 subjects assigned in a 2:1 ratio to test or control lens bilaterally, respectively. Subjects must be otherwise healthy, with myopia between -1.00 D and -6.00 D and astigmatism no greater than 1.00 D that does not interfere with VA.

At the Screening Visit, approximately two-thirds of the eligible subjects will be randomized to receive the test lens (Deseyne [vifilcon C] lenses) and the other one-third eligible subjects will be randomized to receive the control lens (1-Day Acuvue Moist [etafilcon A] lenses). At the Dispensing Visit (Visit 2), subjects will be provided with test or control lenses as part of the dispensing package, along with instructions for the use and care of the lenses. They will be recommended unpreserved lubricating/rewetting solution for use as needed during the study.

Subjects will wear their assigned lenses bilaterally on a daily wear basis, for a minimum of 6 hours/day throughout the study (no maximum time is mandated, as long as subjects do not sleep in their lenses), with additional visits planned for 1 Week (Visit 3), 1 Month (Visit 4), 2 Months (Visit 5), and 3 Months/Exit Visit (Visit 6).

This study follows United States Food and Drug Administration (FDA) Premarket Notification 510(k) Guidance for Daily Wear Contact Lenses adopted in May 1994, and any unpublished subsequent policy declarations.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 40 years of age on the date the informed consent form (ICF) is signed
2. Presence of clear central corneas and absence of any anterior segment disorders in each eye
3. Presence of myopia and requirement for lens correction from -1.00 D to -6.00 D in each eye
4. Best-corrected distance visual acuity (BCDVA) of 50 ETDRS letters (0.1 logMAR) or better in each eye
5. Be an adapted soft contact lens wearer in each eye and agree to wear study lenses in each eye on a daily wear basis and not wear a non-study lens for approximately 3 months
6. Able and willing to comply with all treatment and follow-up/study procedures
7. Able to read, understand, and provide written informed consent on the IRB-approved ICF and provide authorization as appropriate for local privacy regulations

Exclusion Criteria:

1. Participation in any drug or device clinical investigation within 2 weeks prior to Screening and/or during the period of study participation
2. Women of childbearing potential (those who are not surgically sterilized or postmenopausal) who meet any of the following conditions:

   1. Currently pregnant
   2. Plans to become pregnant during the study
   3. Currently breastfeeding
3. History of gas permeable lens wear in either eye within 30 days prior to Screening or history of polymethylmethacrylate lens wear in either eye within 3 months prior to Screening
4. Current monovision, multifocal, or toric contact lens wear in either eye
5. In either eye, current nonabsorbable punctal plug or implantation of absorbable punctal plug within 2 to 6 months (depending on type of absorbable plug) prior to Screening, or punctal plug removal within 2 months prior to Screening. Permanent punctal occlusion in 1 or more puncta or nasolacrimal duct obstruction in either eye is excluded
6. Use of any prescription ocular medication throughout the duration of the study. Prescription eyedrops for dry eye disease (eg, Restasis, Xiidra, Cequa, Eysuvis), as well as nasally administered Tyrvaya, must be discontinued 2 weeks prior to Screening and are prohibited throughout the duration of the study Clinical Study Protocol Version 3.0, 26 April 2023 Page 17 of 66 Bruno Vision Care Protocol 22001
7. Use of over-the-counter eyedrops (eg, oxymetazoline, naphazoline, ketotifen, etc.), except for unpreserved lubricant eyedrops or artificial tears (eg, Systane, Refresh), within 1 week prior to Screening and throughout the duration of the study
8. Use of any systemic or topical medications that may, in the Investigator's opinion, affect ocular physiology or lens performance
9. Anisometropia (spherical equivalent) >2.00 D
10. Ocular astigmatism >1.00 D in either eye
11. Amblyopia in either eye
12. Aphakia in either eye
13. Active ocular disease (eg, dry eye disease, blepharitis, conjunctivitis, keratitis, etc.) in either eye. Subjects must be symptom free for at least 7 days
14. History or evidence of ocular infection within 30 days prior to Screening
15. History or evidence of ocular herpes simplex or ocular herpes zoster
16. Any grade corneal infiltrates in either eye
17. Grade ≥2 finding in either eye during slit lamp examination
18. Any "Present" finding in either eye during slit lamp examination that, in the Investigator's opinion, may interfere with contact lens wear
19. Any scar or neovascularization within the central 4 mm of the cornea in either eye. Subjects with minor peripheral corneal scarring (not extending into the central area) that, in the Investigator's opinion, does not interfere with contact lens wear are eligible to participate in this study
20. History of any corneal surgery (eg, refractive surgery or therapeutic) in either eye
21. Any systemic disease currently affecting ocular health or which, in the Investigator's opinion, may have an effect on ocular health in either eye during the course of the study
22. Allergy to any component in the study care products
23. Meet any of the following criteria:

    1. Subject is an employee of the investigative site
    2. Subject or a member of the subject's household is an ophthalmologist, an optometrist, an optician, or an ophthalmic assistant/technician
    3. Subject or a member of the subject's household is an employee of a manufacturer of contact lenses or contact lens care products
    4. Subject or a member of the subject's household is an employee of a market research firm -

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Slonim, MD, Study Director — iuvobioscience
Locations (3):
- United States (3):
  - Omega Vision Center PA, Longwood, Florida
  - Kennaar Eye Care, Pittsburg, Kansas
  - West Bay Eye Associates, Warwick, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 81 subjects enrolled in the study for a period of 3 months follow-up. Study began on April 8, 2023 at three clinical sites and was completed on January 8, 2024. All sites were at private clinical optometric sites.. Each site conducted screening evaluation to determine eligibility for continuation in the study. Follow-up visits were scheduled at 1 week, 1 month, 2 months, and 3 months including he exit visit. Subjects were instructed to wear the contact lenses a minimum of 6 hours per day.
Pre-assignment Details: The study was designed as a randomized enrollment dictated by an electronic randomization program to test and control. This assignment took place at the screening visit at each site. All subjects were subject to review for inclusion and exclusion at enrollment screening visit. To be included/excluded all screening needed to meet all criteria by forced choice selection. Any positive exclusion element excluded the subject from continuing with participation.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Test Lens. Deseyne Daily Disposable Contact Lens | Control Lens. 1-Day Acuvue Moist Daily Disposable Contact Lens
Started | 53; 106 eyes | 28; 56 eyes
Completed | 53; 106 eyes (The number of subjects required to meet the milestone at study completion was 40 subjects (80 eyes) for the test arm.) | 25; 50 eyes (20 (40 eyes) subjects in the control group to meet milestone at completion of study.)
Not Completed | 0; 0 eyes | 3; 6 eyes
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Lens. Deseyne Daily Disposable Contact Lens | Control Lens. 1-Day Acuvue Moist Daily Disposable Contact Lens | Total
Number analyzed (Participants) | 53 | 28 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 28 | 81
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 18 | 57
  Male | 14 | 10 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 47 | 23 | 70
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 53 | 28 | 81

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Each Post-Baseline Visit in Distance logMAR Visual Acuity (Letters Read) by Eye
Description: To assess each eye for the change from baseline to each post-baseline visit in distance logMAR VA (letters read)
Time Frame: Baseline, Day 1, Week 1, Month 1, Month 2, Month 3
Population: Each row refers to either right eyes (OD) or left eyes (OS); therefore, the number of eyes analyzed is one-half of the total eyes in the study.
Measure: Mean (Standard Deviation); unit: letters read
Units Other Than Participants: eyes
Arm/Group | Test Lens. Deseyne Daily Disposable Contact Lens | Control Lens. 1-Day Acuvue Moist Daily Disposable Contact Lens
Number analyzed (Participants) | 53 | 28
Number analyzed (eyes) | 106 | 56
letters read
  Change from baseline at Day 1 OD: number analyzed (eyes) | 53 | 28
  Change from baseline at Day 1 OD | 0.3 (2.76) | 0.0 (2.47)
  Change from baseline at Week 1 OD: number analyzed (eyes) | 53 | 28
  Change from baseline at Week 1 OD | 0.4 (2.55) | 0.4 (1.94)
  Change from baseline at Month 1 OD: number analyzed (eyes) | 53 | 28
  Change from baseline at Month 1 OD | 0.5 (2.71) | 0.4 (2.83)
  Change from baseline at Month 2 OD: number analyzed (eyes) | 53 | 28
  Change from baseline at Month 2 OD | 0.7 (2.85) | 0.5 (2.38)
  Change from baseline at Month 3 OD: number analyzed (eyes) | 53 | 28
  Change from baseline at Month 3 OD | 0.3 (3.14) | -0.4 (2.81)
  Change from baseline at Day 1 OS: number analyzed (eyes) | 53 | 28
  Change from baseline at Day 1 OS | -0.0 (2.19) | 0.2 (2.56)
  Change from baseline at Week 1 OS: number analyzed (eyes) | 53 | 28
  Change from baseline at Week 1 OS | -0.1 (2.79) | 0.5 (2.12)
  Change from baseline at Month 1 OS: number analyzed (eyes) | 53 | 28
  Change from baseline at Month 1 OS | 0.3 (2.17) | 0.4 (2.86)
  Change from baseline at Month 2 OS: number analyzed (eyes) | 53 | 28
  Change from baseline at Month 2 OS | 0.3 (2.70) | 0.8 (2.58)
  Change from baseline at Month 3 OS: number analyzed (eyes) | 53 | 28
  Change from baseline at Month 3 OS | -0.1 (2.84) | 0.5 (2.52)

2. Primary Outcome: Number and Percentage of Subjects With No More Than 5 Letters Read Loss From Baseline
Description: To assess the number and percentage of subjects with no more than 5 letters read loss from baseline
Time Frame: Day 1, Week 1, Month 1, Month 2, Month 3
Measure: Number; unit: percentage of subjects
Arm/Group | Test Lens. Deseyne Daily Disposable Contact Lens | Control Lens. 1-Day Acuvue Moist Daily Disposable Contact Lens
Number analyzed (Participants) | 53 | 28
percentage of subjects
  Day 1 OD | 98.1 | 100
  Week 1 OD | 100 | 100
  Month 1 OD | 98.1 | 96.0
  Month 2 OD | 98.1 | 100
  Month 3 OD | 94.3 | 96.0
  Day 1 OS | 100 | 96.2
  Week 1 OS | 98.1 | 100
  Month 1 OS | 100 | 96.0
  Month 2 OS | 100 | 96.0
  Month 3 OS | 98.1 | 96.0

3. Primary Outcome: Slit Lamp Findings Grade >2 at Any Follow-Up Visit
Description: To assess the following slit lamp findings: epithelial edema, epithelial microcysts, limbal injection, bulbar injection, upper lid tarsal conjunctival, corneal neovascularization, and corneal infiltrates
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Test Lens. Deseyne Daily Disposable Contact Lens | Control Lens. 1-Day Acuvue Moist Daily Disposable Contact Lens
Number analyzed (Participants) | 53 | 26
Participants
  Any slit lamp findings Grade >2 | 0 | 0
  No slit lamp findings Grade >2 | 53 | 26

4. Secondary Outcome: Symptoms/Complaints
Description: This unnamed questionnaire measures change from baseline in discomfort, excessive tearing, photophobia, halos, itching/burning/spectacle blur, variable vision, blurred vision, lens needs cleaning, handling using a 0 (no symptoms) to 4 (severe symptoms) scale for each symptom
Time Frame: Month 3
Population: Each row analyzes either right eyes (OD) or left eyes (OS); therefore, the number of eyes analyzed is one-half of the total eye population in that arm
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Test Lens. Deseyne Daily Disposable Contact Lens | Control Lens. 1-Day Acuvue Moist Daily Disposable Contact Lens
Number analyzed (Participants) | 53 | 28
Number analyzed (eyes) | 106 | 56
units on a scale
  Change from baseline in discomfort OD: number analyzed (eyes) | 53 | 28
  Change from baseline in discomfort OD | 0.6 (0.80) | 0.4 (0.96)
  Change from baseline in discomfort OS: number analyzed (eyes) | 53 | 28
  Change from baseline in discomfort OS | 0.6 (0.79) | 0.4 (0.96)
  Change from baseline in excessive tearing OD: number analyzed (eyes) | 53 | 28
  Change from baseline in excessive tearing OD | 0.0 (0.00) | 0.0 (0.00)
  Change from baseline in excessive tearing OS: number analyzed (eyes) | 53 | 28
  Change from baseline in excessive tearing OS | 0.0 (0.00) | 0.0 (0.00)
  Change from baseline in photophobia OD: number analyzed (eyes) | 53 | 28
  Change from baseline in photophobia OD | 0.0 (0.00) | -0.1 (0.40)
  Change from baseline in photophobia OS: number analyzed (eyes) | 53 | 28
  Change from baseline in photophobia OS | 0.0 (0.00) | -0.1 (0.41)
  Change from baseline in halos OD: number analyzed (eyes) | 53 | 28
  Change from baseline in halos OD | 0.0 (0.00) | -0.1 (0.40)
  Change from baseline in halos OS: number analyzed (eyes) | 53 | 28
  Change from baseline in halos OS | 0.0 (0.00) | -0.1 (0.41)
  Change from baseline in itching/burning OD: number analyzed (eyes) | 53 | 28
  Change from baseline in itching/burning OD | -0.0 (0.50) | 0.1 (0.40)
  Change from baseline in itching/burning OS: number analyzed (eyes) | 53 | 28
  Change from baseline in itching/burning OS | 0.0 (0.52) | 0.1 (0.50)
  Change from baseline in spectacle blur OD: number analyzed (eyes) | 53 | 28
  Change from baseline in spectacle blur OD | 0.0 (0.00) | 0.0 (0.00)
  Change from baseline in spectacle blur OS: number analyzed (eyes) | 53 | 28
  Change from baseline in spectacle blur OS | 0.0 (0.00) | 0.0 (0.00)
  Change from baseline in variable vision OD: number analyzed (eyes) | 53 | 28
  Change from baseline in variable vision OD | 0.1 (0.45) | 0.1 (0.28)
  Change from baseline in variable vision OS: number analyzed (eyes) | 53 | 28
  Change from baseline in variable vision OS | 0.1 (0.45) | 0.1 (0.28)
  Change from baseline in blurred vision OD: number analyzed (eyes) | 53 | 28
  Change from baseline in blurred vision OD | 0.0 (0.19) | 0.2 (0.62)
  Change from baseline in blurred vision OS: number analyzed (eyes) | 53 | 28
  Change from baseline in blurred vision OS | 0.1 (0.33) | 0.2 (0.62)
  Change from baseline in lens needs cleaning OD: number analyzed (eyes) | 53 | 28
  Change from baseline in lens needs cleaning OD | 0.0 (0.19) | -0.0 (0.20)
  Change from baseline in lens needs cleaning OS: number analyzed (eyes) | 53 | 28
  Change from baseline in lens needs cleaning OS | 0.0 (0.19) | -0.0 (0.20)
  Change from baseline in handling OD: number analyzed (eyes) | 53 | 28
  Change from baseline in handling OD | 0.5 (1.07) | 0.4 (0.87)
  Change from baseline in handling OS: number analyzed (eyes) | 53 | 28
  Change from baseline in handling OS | 0.6 (1.05) | 0.5 (0.88)

5. Secondary Outcome: Lens Wettability, Centration, and Movement
Description: Wettability Analog Scale 0-4 (0=100% wettable, 4=more than one dry spot greater than 0.5 mm) Lower score is better Centration Analog Scale 0-4 (0=superior cornea, 4=inferior cornea) Lower score is better Movement Analog Scale 0-4 (0=adequate, 4=adherence to cornea) Lower score is better
Time Frame: 3 months
Population: Each row analyzes either right eyes (OS) or left eyes (OS); therefore, the total number of eyes in a row is one-half of the total eye population for that arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Test Lens. Deseyne Daily Disposable Contact Lens | Control Lens. 1-Day Acuvue Moist Daily Disposable Contact Lens
Number analyzed (Participants) | 53 | 28
Number analyzed (eyes) | 106 | 56
units on a scale
  Change from baseline in wettability OD: number analyzed (eyes) | 53 | 28
  Change from baseline in wettability OD | 0.1 (0.32) | 0.1 (0.33)
  Change from baseline in wettability OS: number analyzed (eyes) | 53 | 28
  Change from baseline in wettability OS | 0.1 (0.32) | 0.1 (0.28)
  Change from baseline in centration OD: number analyzed (eyes) | 53 | 28
  Change from baseline in centration OD | 0.1 (0.36) | 0.0 (0.61)
  Change from baseline in centration OS: number analyzed (eyes) | 53 | 28
  Change from baseline in centration OS | 0.1 (0.40) | 0.0 (0.73)
  Change from baseline in movement OD: number analyzed (eyes) | 53 | 28
  Change from baseline in movement OD | 0.0 (0.39) | 0.0 (0.35)
  Change from baseline in movement OS: number analyzed (eyes) | 53 | 28
  Change from baseline in movement OS | 0.1 (0.45) | 0.0 (0.35)

6. Secondary Outcome: Lens Deposits
Description: To assess type of deposit
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Test Lens. Deseyne Daily Disposable Contact Lens | Control Lens. 1-Day Acuvue Moist Daily Disposable Contact Lens
Number analyzed (Participants) | 53 | 25
Participants
  No deposits | 51 | 22
  Film | 0 | 1
  Spots | 2 | 2

ADVERSE EVENTS:
Time Frame: 3 months
Description: Treatment-emergent adverse events using system organ class and preferred terms
Arm/Group | Test Lens. Deseyne Daily Disposable Contact Lens | Control Lens. 1-Day Acuvue Moist Daily Disposable Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/26
Other Adverse Events (participants affected / at risk) | 3/53 | 1/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Lens. Deseyne Daily Disposable Contact Lens (N=53) | Control Lens. 1-Day Acuvue Moist Daily Disposable Contact Lens (N=26)
Contact lens intolerance (Eye disorders) | 0 (0) | 1 (2)
Vision blurred (Eye disorders) | 0 (0) | 1 (2)
Hordeolum (Eye disorders) | 1 (1) | 0 (0)
Lacrimation decreased (Eye disorders) | 1 (1) | 0 (0)
Vital dye staining cornea present (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication or presentation, a copy of the final text should be forwarded by the Investigator(s) to the Sponsor or its designee, for comment. Such comments shall aim to ensure the scientific integrity of the proposed publications and/or presentations and ensure that the data and material referring to Sponsor products and activities receive fair, accurate, and reasonable presentation.

DOCUMENTS (2):
  • Study Protocol (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT05927753/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT05927753/SAP_001.pdf